CLINICAL TRIAL: NCT06922201
Title: SUstaiNable inteRventions and Healthy behavIours for adoleScent Primary prEvention of Cancer With Digital Tools. Study 1: SmartCoach
Brief Title: The SUNRISE Project is Dedicated to Enhancing Primary Cancer Prevention Among Adolescents in Europe by Leveraging Innovative Digital Tools and Methodologies. SmartCoach, Developed by Swiss Research Institute for Public Health and Addiction (ISGF), is a Mobile Phone-based Life-skills Training Program
Acronym: SUNRISE_1
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Biobizkaia Health Research Institute (Other Government)
Collaborators: University Ghent (Other); FEDERAZIONE ITALIANA DELLE ASSOCIAZIONI DI VOLONTARIATO IN ONCOLOGIA (Unknown); Hellenic Mediterranean University (Other); University of Zurich (Other); FISABIO (Foundation for the Promotion of Healthcare and Biomedical Research in the Valencian Community) (Unknown); Cyprus Association of Cancer Patients and Friends (PASYKAF) (Unknown); Alma Mater Europaea University (Unknown); The Oncology Institute "Prof. Dr. Ion Chiricuţă" Cluj-Napoca (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SUNRISE_Study1
Record Dates: First submitted 2024-12-05; First posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2024-12

CONDITIONS: Cancer
Keywords: SUNRISE; SmartCoach; Life-skills training; substance use prevention; adolescents
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Prospective, multicentre, multinational, 2-arm, parallel-group, hybrid effectiveness implementation cluster randomized control trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): No intervention
- Intervention (Experimental): SmartCoach program
  Interventions: Other: SmartCoach

INTERVENTIONS:
Other: SmartCoach — Participants will receive a tailored life-skills training program over four months, which includes 2-4 personalized messages per week via Whatsapp. These messages, in the form of microdialogues generated by an automated system, will focus on self-management skills, social skills and substance use resistance skills. The program will use interactive elements such as quiz questions, behavioural plans, message contests and multimedia content (audio testimonials, motivational podcasts, videos, images and links to relevant websites).
  Arms: Intervention

SUMMARY:
SUNRISE aims to create a comprehensive, engaging, and sustainable digital health promotion program that not only addresses immediate health behaviours but also instills lifelong healthy habits among adolescents. By integrating cutting-edge digital tools with traditional educational settings, SUNRISE seeks to bridge the gap between knowledge and practice, making cancer prevention a tangible and achievable goal for young people. This study represents a significant step towards reducing the future burden of cancer through early and innovative preventive measures.

The SUNRISE project aims to test its intervention on students across eight European countries, including Greece, Switzerland, Slovenia, Spain, Cyprus, Italy, Belgium, and Romania. This study focuses on integrating digitally enhanced programs into the school environment, targeting students aged 10 to 19 years. The program emphasizes inclusivity, ensuring participation from both urban and rural regions and socially disadvantaged groups such as ethnic minorities and migrants. By addressing diverse socio-economic, cultural, and environmental contexts, SUNRISE aspires to create a universally applicable and impactful intervention.

Specifically, this study is focus on the SmartCoach program, developed by the Swiss Research Institute for Public Health and Addiction (ISGF). It is a mobile phone-based life-skills training program designed to prevent substance use among adolescents. It will integrate digital tools and leveraging social media creating a more engaging, effective and sustainable intervention for adolescent health behaviour change.

The SmartCoach solution will be significantly more effective than an assessment-only approach in preventing the initiation and escalation of problematic alcohol and tobacco use. This efficacy will be demonstrated through a two-arm cluster-randomized controlled trial, with participants assessed at baseline, 6 months, and 18 months. The study will measure key outcomes related to substance use frequencies, intensities, and associated behavioral changes, showing that the individually tailored 4 month intervention program leads to greater reductions in these behaviors compared to the control group over the 18-month follow-up period.

DETAILED DESCRIPTION:
Cancer is a leading cause of death worldwide, responsible for an estimated 9.9 million deaths in 2020. Many cancers can currently be prevented by avoiding risk factors, implementing evidence-based prevention strategies, and adopting healthy behaviours. Adolescence is a critical period for establishing these behaviours, as many risk behaviours such as smoking and poor diet begin at this stage. Despite numerous school-based interventions, significant gaps remain in achieving sustainable health behaviour changes among adolescents.

The SUNRISE project aims to bridge these gaps and reduce social inequalities in primary cancer prevention among adolescents in Europe. Traditional health promotion programs face barriers such as the need for extensive resources and continuous support for educators. Digital interventions offer a promising solution by providing cost-effective, engaging, and tailored content accessible 24/7. As part of its comprehensive approach, SUNRISE seeks to test various innovative solutions, including the SmartCoach program, to determine the most effective strategies for adolescent health promotion.

SmartCoach, developed by Swiss Research Institute for Public Health and Addiction (ISGF), is a mobile phone-based life-skills training program designed to prevent substance use among adolescents. It has shown significant long-term effectiveness in reducing tobacco smoking and cannabis use. Based on Social Cognitive Theory, SmartCoach promotes self-management skills, social skills, and substance use resistance through tailored weekly text messages over a period of several months.

Adolescence is a period of significant biological, psychological, and social transitions. These transitions provide opportunities for skill development but also present risks for developing harmful behaviours. Substance use often begins during adolescence, with increased prevalence of alcohol, tobacco, and cannabis consumption as teen's age. For instance, the Health Behaviour in School-aged Children (HBSC) study showed noticeable increases in the lifetime prevalence of these substances among 11-to-15-year-olds. Schools are ideal settings for delivering preventive interventions due to their accessibility to young people.

Life-skills training programs, which focus on self-management, social skills, and substance use resistance, have proven effective but face challenges in implementation and sustainability. Traditional face-to-face interventions require substantial resources and commitment from educators. Digital interventions, such as those delivered via mobile phones, can overcome these obstacles by providing flexible, engaging, and tailored content.

SmartCoach addresses key concepts of Social Cognitive Theory, such as outcome expectations, self-efficacy, observational learning, facilitation, and self-regulation. The program in its previous version provided:

* Automated Messaging: 2-4 messages per week focusing on self-management skills, social skills, and substance use resistance.
* Interactive Features: Quizzes to tailor behavioural plans, friendly competitions to incentivize engagement, and integration with social media platforms like YouTube.

A cluster-randomized controlled trial in Switzerland showed high acceptance and promising effectiveness of SmartCoach among secondary and upper secondary school students, with significant longer-term reductions in tobacco- and cannabis use prevalence. Active program engagement was stimulated by interactive features such as quiz questions, message and picture contests, and the integration of a friendly competition with prizes, where users collected credits with each interaction.

Popular online social media platforms (e.g., WhatsApp, YouTube, TikTok) play a significant role in young people's lives and offer powerful spaces to reach them and influence their health. These platforms provide interactive functionalities and have great potential for user engagement and retention. Health behaviour change interventions using social media have shown modest evidence of effectiveness, and there have been calls to strengthen research targeting adolescents and the sustainability of their behaviour changes in the longer term. An automated WhatsApp-based coaching program for smoking cessation developed by ISGF provides a foundation for further development within the SUNRISE project.

SmartCoach will be enhanced within the SUNRISE project by leveraging the interactive and engaging features of social media platforms. Adolescents spend a considerable amount of time on platforms like WhatsApp, YouTube, and TikTok, making these platforms ideal for delivering health interventions. By integrating SmartCoach with these social media platforms, the program aims to increase engagement, retention, and effectiveness.

For instance, WhatsApp can be used to send automated messages and provide a communication channel for adolescents to interact with addiction experts. YouTube and TikTok can be used to share engaging multimedia content that promotes healthy behaviours and provides educational resources about cancer prevention. These platforms can also facilitate peer support and create a community of adolescents who are committed to adopting healthier lifestyles.

By integrating digital tools and leveraging social media, SmartCoach aims to create a more engaging, effective, and sustainable intervention for adolescent health behaviour change. The focus is primarily on preventing substance use and promoting healthy lifestyles to reduce the risk of cancer. The SUNRISE project seeks to bridge existing gaps in adolescent health promotion, reduce social inequalities in primary cancer prevention, and become a reference point in Europe and beyond for adolescents, their parents, educators, and public health experts.

The SUNRISE project and the SmartCoach program represent a significant step forward in the primary prevention of cancer among adolescents. By addressing the challenges of traditional health promotion programs and leveraging the power of digital interventions, these initiatives aim to create lasting health behaviour changes that will reduce the risk of cancer and improve overall health outcomes for future generations.

ELIGIBILITY:
Inclusion Criteria:

* Minimum Age: Students must be at least 14 years old at the time of enrolment.
* Mobile Device and Internet Access: Students must have access to a smartphone and the Internet.
* Informed Consent: Students must provide their signed informed consent to participate in the study.
* Parental Consent: Students must obtain and submit signed informed consent from a parent or legal guardian.

Exclusion Criteria:

* Age Restrictions: Students who are younger than 14 years or older than the established age range for participation.
* Consent Issues: Students who have not signed the informed consent form or do not have signed informed consent from their parents or legal guardians.
* Follow-up Limitations: Students who are unable to commit to the follow-up period of at least 18 months or are unlikely to complete the study.

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 3500 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Point prevalence rate of tobacco or nicotine use | The primary outcomes will be assessed at baseline, 6 months, and 18 months follow-up
  This will be measured by assessing the rate of abstinence (not even smoked a puff or used once) from tobacco or nicotine products in the preceding 30 days.

SECONDARY OUTCOMES:
Frequency of tobacco cigarette smoking | The secondary outcomes will also be assessed at baseline, 6 months, and 18 months follow-up
  Determined by the number of days on which tobacco cigarettes were smoked in the last 30 days
Prevalence and frequency of other nicotine products use | The secondary outcomes will also be assessed at baseline, 6 months, and 18 months follow-up
  Determined by the number of days on which other nicotine products, e.g., vape, e-cigarette, e-shisha, snus or nicotine pouches, were consumed in the last 30 days
Prevalence and frequency of cannabis use | The secondary outcomes will also be assessed at baseline, 6 months, and 18 months follow-up
  Measured by the number of cannabis (containing THC) consumption days in the preceding 30 days
Prevalence and frequency of alcohol use | The secondary outcomes will also be assessed at baseline, 6 months, and 18 months follow-up
  Assessed by the number of alcohol use days in the preceding 30 days
Perceived Stress | The secondary outcomes will also be assessed at baseline, 6 months, and 18 months follow-up
  Measured using the 4-item version of the Perceived Stress Scale (PSS-4): The questions in this scale ask about the feelings and thoughts during the last month. In each case, the response represents how often participant felt or thought a certain way.
  Scoring Instructions:
  Total score is determined by adding together the scores of each of the four items. Questions 2 and 3 are reverse coded.
  Questions 1 and 4: 0 = Never; 1 = Almost never; 2 = Sometimes; 3 = Fairly often; 4 = Very often Questions 2 and 3: 4 = Never; 3 = Almost never; 2 = Sometimes; 1 = Fairly often; 0 = Very often Lowest score: 0; Highest score: 16. Higher scores are correlated to more stress.
Social skills | The secondary outcomes will also be assessed at baseline, 6 months, and 18 months follow-up
  Assessed utilizing the brief version of the Interpersonal Competence Questionnaire-10 (ICQ-10), which encompasses the following 5 domains: (1) initiation of relationships, (2) negative assertions, (3) disclosure of personal information, (4) emotional support, and (5) conflict management.
  Scoring instructions: Good=4; Fairly good= 3; Rather poor=2; Poor=1. Total score is determined by adding the value of all items and dividing by 2. Maximum value= 20; Minimum value= 5. The higher the score, the higher the interpersonal competence.
Healthy eating habits | The secondary outcomes will also be assessed at baseline, 6 months, and 18 months follow-up
  Measured using the WHO/HBSC eating habits questionnaire. Label values: 1 = never, 2 = Less than once a week, 3 = Once a week, 4 = 2-4 days a week, 5 = 5-6 days a week, 6 = Once a day (Every day), 7 = Every Day (more than once).
EuroQoL-5D-5L questionnaire | The secondary outcomes will also be assessed at baseline, 6 months, and 18 months follow-up
  Scoring from 0-100 points. 0 points low quality of life 100 high quality of life

CONTACTS AND LOCATIONS:
Locations (8):
- Ghent University (UGENT), Ghent, Belgium
- Cyprus Association of Cancer Patients and Friends (PASYKAF), Nicosia, Cyprus
- Hellenic Mediterranean University (HMU), Heraklion, Greece
- Italian Federation of Voluntary Associations in Oncology (FAVO), Roma, Italy
- Institute of Oncology "Prof dr. Ion Chiricuta" CLUJ NAPOCA (IOCN), Cluj-Napoca, Romania
- Alma Mater Europaea University (AMEU), Maribor, Slovenia
- Foundation for the Promotion of Health and Biomedical Research of the Valencian Community (Fisabio, Valencia, Spain
- Swiss Research Institute for Public Health and Addiction (ISGF), Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maher CA, Lewis LK, Ferrar K, Marshall S, De Bourdeaudhuij I, Vandelanotte C. Are health behavior change interventions that use online social networks effective? A systematic review. J Med Internet Res. 2014 Feb 14;16(2):e40. doi: 10.2196/jmir.2952. PMID 24550083
- [Background] Bandura A. Health promotion by social cognitive means. Health Educ Behav. 2004 Apr;31(2):143-64. doi: 10.1177/1090198104263660. PMID 15090118
- [Background] Haug S, Schaub MP, Venzin V, Meyer C, John U. Efficacy of a text message-based smoking cessation intervention for young people: a cluster randomized controlled trial. J Med Internet Res. 2013 Aug 16;15(8):e171. doi: 10.2196/jmir.2636. PMID 23956024
- [Background] Stockings E, Hall WD, Lynskey M, Morley KI, Reavley N, Strang J, Patton G, Degenhardt L. Prevention, early intervention, harm reduction, and treatment of substance use in young people. Lancet Psychiatry. 2016 Mar;3(3):280-96. doi: 10.1016/S2215-0366(16)00002-X. Epub 2016 Feb 18. PMID 26905481
- [Background] Thomas RE, McLellan J, Perera R. School-based programmes for preventing smoking. Cochrane Database Syst Rev. 2013 Apr 30;2013(4):CD001293. doi: 10.1002/14651858.CD001293.pub3. PMID 23633306
- [Background] Haug S, Paz Castro R, Wenger A, Schaub MP. A Mobile Phone-Based Life-Skills Training Program for Substance Use Prevention Among Adolescents: Cluster-Randomized Controlled Trial. JMIR Mhealth Uhealth. 2021 Jul 13;9(7):e26951. doi: 10.2196/26951. PMID 34255703
- [Background] Champion KE, Parmenter B, McGowan C, Spring B, Wafford QE, Gardner LA, Thornton L, McBride N, Barrett EL, Teesson M, Newton NC; Health4Life team. Effectiveness of school-based eHealth interventions to prevent multiple lifestyle risk behaviours among adolescents: a systematic review and meta-analysis. Lancet Digit Health. 2019 Sep;1(5):e206-e221. doi: 10.1016/S2589-7500(19)30088-3. Epub 2019 Aug 19. PMID 33323269
- [Background] Paz Castro R, Haug S, Wenger A, Schaub MP. Longer-Term Efficacy of a Digital Life-Skills Training for Substance Use Prevention. Am J Prev Med. 2022 Dec;63(6):944-953. doi: 10.1016/j.amepre.2022.06.017. Epub 2022 Aug 18. PMID 35985899
- [Background] Domitrovich CE, Durlak JA, Staley KC, Weissberg RP. Social-Emotional Competence: An Essential Factor for Promoting Positive Adjustment and Reducing Risk in School Children. Child Dev. 2017 Mar;88(2):408-416. doi: 10.1111/cdev.12739. Epub 2017 Feb 18. PMID 28213889
- [Background] Al-Hosni K, Chan MF, Al-Azri M. The Effectiveness of Interventional Cancer Education Programs for School Students Aged 8-19 Years: a Systematic Review. J Cancer Educ. 2021 Apr;36(2):229-239. doi: 10.1007/s13187-020-01868-1. PMID 32895878
- [Background] Herlitz L, MacIntyre H, Osborn T, Bonell C. The sustainability of public health interventions in schools: a systematic review. Implement Sci. 2020 Jan 6;15(1):4. doi: 10.1186/s13012-019-0961-8. PMID 31906983
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- See also: HBSC- Health Behaviour School-aged Cildren — https://data-browser.hbsc.org/